CLINICAL TRIAL: NCT07025096
Title: Evaluating Artificial Intelligence-Based Comprehensive Clinical Decision Support for Sepsis and ARDS
Brief Title: Evaluating Artificial Intelligence-Based Clinical Decision Support for Sepsis and ARDS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 858201; R35GM155262 (NIH)
Record Dates: First submitted 2025-05-30; First posted 2025-06-17 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Sepsis; Acute Respiratory Distress Syndrome (ARDS)
Keywords: Sepsis; Acute Respiratory Distress Syndrome; Clinical Decision Support; Clinical Decision Support System; Invasive Mechanical Ventilation; Artificial Intelligence
MeSH Terms: conditions — Sepsis; Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will review a series of clinical vignettes. Each vignette will be randomized to show a treatment recommendation either from an artificial intelligence-based clinical decision support system (AI CDSS) or from the clinician in the case, reflecting actual clinical practice. Vignettes will be randomized equally, and participants will see an equal number of vignettes from each arm.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial Intelligence (Experimental): Critical care cases / vignettes in this arm will contain treatment recommendations generated by an artificial intelligence-based clinical decision support system. Each participant will review four vignettes from this arm.
  Interventions: Other: Artifical Intelligence-Generated Treatment Recommendations
- Human Clinician (No Intervention): Critical care cases / vignettes in this arm will contain treatment recommendations that were enacted by the clinician in the actual case. Each participant will review four vignettes from this arm.

INTERVENTIONS:
Other: Artifical Intelligence-Generated Treatment Recommendations — The clinical vignette will contain treatment recommendations which were generated by an artificial intelligence-based clinical decision support system.
  Arms: Artificial Intelligence

SUMMARY:
Sepsis and acute respiratory distress syndrome (ARDS) are common in intensive care units. Managing sepsis and ARDS is inherently complex and requires making numerous decisions under uncertainty. Artificial intelligence (AI) clinical decision support systems (CDSSs) offer a promising approach to support care management for sepsis and ARDS.

The goal of this randomized, survey-based study is to compare treatment recommendations enacted by clinicians to those generated by an AI CDSS. The study will investigate whether an AI CDSS can generate treatment recommendations that are safe, appropriate, and indistinguishable to those provided by real clinicians.

In this study, participants (i.e., critical care clinicians) will review a series of critical care cases (vignettes) in an electronic survey. Each vignette will contain a de-identified case of a patient with sepsis and ARDS as well as treatment recommendations for the case. Participants will assess the safety and appropriateness of each treatment recommendations and answer whether they think the treatment recommendations came from the clinician or an AI CDSS.

ELIGIBILITY:
Inclusion Criteria:

* Working as a physician (i.e., MD, DO) or an advanced practice provider (i.e., nurse practitioner, physician assistant)
* Working at a hospital or medical center in medical critical care, anesthesia critical care, surgical critical care, or emergency medicine

Exclusion Criteria:

* Has not completed a residency training program (i.e., medical intern or resident)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Predicting the Source of Treatment Recommendation | From enrollment to the end of the survey, an average of 45 minutes
  Participants will answer if they think the treatment recommendations came from artificial intelligence (AI) or a clinician for each clinical vignette. Accuracy will be measured by participants correctly identifying the source of treatment recommendation.

SECONDARY OUTCOMES:
Confidence of Predicting the Source of Treatment Recommendation | From enrollment to the end of the survey, an average of 45 minutes
  Participants will respond to their confidence in their prediction in whether the treatment recommendations of a vignette came from artificial intelligence or from a clinician. Confidence will measured on a Likert scale ranging from 0 (Not at all confident) to 7 (Extremely confident).
Appropriateness of Treatment Recommendations | From enrollment to the end of the survey, an average of 45 minutes
  Appropriateness will be measured by participants' assessments of the clinical appropriateness of the treatment recommendations in the vignettes via Yes-No and free-text responses.
Safety of Treatment Recommendations | From enrollment to the end of the survey, an average of 45 minutes
  Safety will be measured by participants' assessments of the overall safety of the treatment recommendations in the vignettes via Yes-No and free-text responses.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Weissman, MD, MSHP, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Angeli Gazola A, Bishop NS, Schmid BE, Pirracchio R, Valley TS, Bhavani SV, Krutsinger DC, Giannini HM, Lu Y, Ungar LH, Meyer NJ, Kerlin MP, Weissman GE. Evaluating AI-based comprehensive clinical decision support for sepsis and ARDS: protocol for a Clinician Turing Test. BMJ Open. 2025 Dec 24;15(12):e106757. doi: 10.1136/bmjopen-2025-106757. PMID 41448698